CLINICAL TRIAL: NCT07015099
Title: Delayed Transfer to Spinal Injury Unit Post Acute Traumatic Spinal Cord Injury: A Comprehensive Assessment on Health Impacts and Rehabilitation
Brief Title: Complications Associated With Delayed Admission to Spinal Injury Unit
Status: Not yet recruiting | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1 917
Record Dates: First submitted 2025-05-14; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injury; Delayed Admission
Keywords: SCI; Spinal Cord Injury; Delayed admission
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine the prevalence of complications including PUs at time of admission to a regional spinal injury rehabilitation unit (MCSI), the relationship between wait time to admission for specialist SCI rehabilitation and complication n occurrence, neurological recovery, and length of stay. The hypothesis is that wait time to transfer from the acute hospital to the specialised SCI rehabilitation unit is associated with increased PU prevalence and other SCI complications, as well as poorer neurological recovery and increased length of stay.

DETAILED DESCRIPTION:
Pressure ulcers (PUs) are one of many challenging complications in patients with spinal cord injury (SCI). PUs impact on length of rehabilitation, activities of daily living, participation in physical and social activities, health-related quality of life and increases health care costs significantly. Globally, approximately 32% of patients with SCI experience PUs and this may reflect inadequate prevention and management strategies.

Complications including PUs can occur at any time following SCI from the acute phase, the rehabilitation phase and during the long term follow up period, however the highest PU risk is in the acute phase. Older age, decreased general health status and prolonged periods of immobilisation increases risk of PUs in the acute period. Specialised SCI rehabilitation centres are recommended to reduce the overall length of stay (LOS), mortality and reduce complications following SCI.

Variations exist globally between time to admission for specialist rehabilitation from onset of acute traumatic spinal cord injury with averages of 7.3-377 days reported in the literature. Some identified barriers to specialised SCI rehabilitation unit admission include lack of bed availability, shortage of skilled staff, inadequate finance, physical and environmental barriers resulting in increased wait times for specialist rehabilitation. Time to admission to specialist rehabilitation unit greater than one month have been shown to increase the occurrence of complications, including PUs at the time of rehabilitation admission.

A review conducted in 2003 by Bagnall et al., evaluated 22 articles which compared early admission to a specialist SCI unit to late admission and/or no admission. Whilst favourable neurological recovery was suggested for those who were admitted to a specialist centre compared to late or no admission, all the studies included in the review were deemed to be of poor quality, conducted in the 1980/1990s and, in most cases, could not separate the time of referral to an SCI centre to the time of admission.

In 2015, the All Party Parliamentary Group on SCI undertook an inquiry into the impact of nationwide SCI centres and the people they support. They reported that from 118 patients waiting for admission to a SCI unit, contact with an SCI unit on the same day as the injury was only made for 9 patients. The median time from injury to contact with a specialist centre was 6 days and the median time from injury to referral to a SCI centre was 8 days. On further investigation, 36% of cases required additional information before admission suitability, 24% of cases were due to bed availability, 20% of cases were accepted but were later deemed clinically unfit for transfer, 10% were deemed suitable for outreach or out-patient services and the final 10% of cases were deemed 'other'.

However, this is not the case in every part of the UK. In a recent 2023/24 report from The Queen Elizabeth National Spinal Injuries Unit (Glasgow), it was stated that there was no waiting list for admission to the SCI unit for that period, and of those patients referred to the centre, 58% of patients were admitted within one week. It was reported that the mean admission time to the SCI unit was 29 days, compared to the mean admission time for other spinal centres in the UK being 2-3 months.

The effect of delayed admission to a SCI centre for both the individual with injury and the surrounding family can be profound. Not only are patients often in a high state of uncertainty about their possible prognosis but they can also feel extremely overwhelmed by all the unanswered questions. For those who are waiting to be admitted to a SCI unit, a fear of losing their 'window of opportunity', of which may potentially alter their expected functional recovery, can be seen amongst the patients, highlighted in the evidence above. Delayed admission can also lead to a heightened risk of complications such as PUs, contractures and infections, secondary to an increased hospital stay and decreased functional recovery.

An initial service evaluation from January 2016 and December 2018 has been undertaken by clinicians on the MCSI (RJAH) in the last year to begin to investigate the impact of delayed referral to the MCSI on the prevalence of PUs, it found via multivariate analysis that age, sex and wait time to admission for specialist SCI rehabilitation were significant risk factors for the development of PUs. Here it is proposed to build on this study by undertaking a comprehensive analysis using the last decade of data, to evaluate the impact of delayed admission on SCI rehabilitation and neurological recovery.

ELIGIBILITY:
Inclusion Criteria:

All eligible patients will be included, of both sexes.

Exclusion Criteria:

Patients younger than 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be included if they were 18 years or older at the time of the injury and admitted to MCSI and had an SCI classified by the American Spinal Injury Association Impairment Scale (ASIA) A-D.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Relationship between wait time to admission and complications | 7 months
  Descriptive statistics and hypothesis-testing methods will be used to analyse primary data. Central tendencies (arithmetic mean, median and frequencies) and measures of variability (standard deviation and interquartile ranges) will be obtained. To test the hypothesis of the difference in frequency (sex) and difference in arithmetic means (age), chi-squared test and t-test will be used respectively. Mann-Whitney U-test will be used to test the hypothesis of difference in wait time to transfer for specialist SCI rehabilitation. Multivariable linear and generalised linear regression will be undertaken to identify the potential predictors associated with complication risk, patient recovery and hospital stay from delayed admission to the MCSI rehabilitation centre.

CONTACTS AND LOCATIONS:
Locations (1):
- The Robert Jones and Agnes Hunt Orthopaedic Hospital, Oswestry, United Kingdom

IPD SHARING:
Plan to Share IPD: No